CLINICAL TRIAL: NCT04705233
Title: A 2 Arm, Multi-centre, Open Label, Parallel-group Randomised Designed Trial Investigating the Use of Sputum Colour Charts to Guide Antibiotic Self-treatment of Acute Exacerbation of COPD in Patients With COPD - Colour COPD
Brief Title: Sputum Colour Charts to Guide Antibiotic Self-treatment of Acute Exacerbation of COPD (Colour COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Salford Royal Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RG_18-088
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Airflow Obstruction,; Chronic COAD; COPD; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; Primary Care; Primary Healthcare; Patient Care; Chronic Bronchitis; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: A 2 arm, multi-centre, open label, parallel-group randomised designed trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sputum chart (Experimental): Use of the 5 point sputum colour chart, adapted from Bronkotest® a self-management (SM) plan and rescue pack (RP) containing 5 days supply of antibiotic and steroid treatment
  Interventions: Other: sputum colour chart
- Control (No Intervention): Use of the plan and rescue pack alone (best usual care)

INTERVENTIONS:
Other: sputum colour chart — 5-point Sputum Colour Chart plus best standard care
  Arms: Sputum chart

SUMMARY:
The primary objective of this study is to determine if a sputum colour chart can aid patient self-management of COPD exacerbations, such that use of the chart is non-inferior to usual care with respect to hospital admissions. There are also a range of other secondary objectives as detailed in the secondary outcomes section. An integral pilot phase, economic evaluation and process evaluation are also included.

DETAILED DESCRIPTION:
This study is a pragmatic, individually randomized trial, set in primary care, comparing usual care to the use of a sputum colour chart in patients at risk of hospital admission for Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD), with the hypothesis that use of a colour chart will be non-inferior to usual care with respect to hospital admission rate after 12 months of follow-up, this being the primary outcome measure. Use of a chart might reduce antibiotic use, and thus might also change patterns of antibiotic resistance long term, such that these are important secondary outcomes. There is an internal pilot phase, a detailed process evaluation and a cost-effectiveness study.

The trial protocol also includes three sub-studies: 1) using a daily electronic symptom diary capable of picking up symptom defined (but potentially unreported) AECOPD, since these are an important prognostic marker (section 3); 2) collecting sputum samples from patients to assess patterns of antibiotic resistance and 3) a qualitative study which will include staff (for example, healthcare staff delivering the intervention) and patients.

This trial uses a sputum colour chart as part of a self-management intervention that enables patients with COPD to determine whether they have an exacerbation, and whether this requires antibiotic treatment. The 5 point sputum colour chart, adapted from Bronkotest® is being used.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed COPD, confirmed by a medical record of post-bronchodilator spirometry denoting obstruction.
* ≥2 AECOPD in the 12 months prior to screening according to the patient or ≥1 hospital admission for AECOPD (i.e. Global Initiative for Chronic Obstructive Lung Disease- GOLD; C or D).
* Able to safely use SM plan in the view of their usual care practitioner
* Able to use sputum colour chart; this will be confirmed by a sight test if there is any doubt on initial assessment by the usual care or research team. Patients who report being colour blind will have their ability to use the chart tested at the screening visit.
* Written Informed consent given

Additionally, to participate in the E-diary sub-study. - Access to smartphone/tablet and an email address.

Additionally, to participate in the Sputum sub-study.

- Chronic bronchitis, defined by self-reported sputum production for at least 3 months in each of 2 consecutive years or more.

Exclusion Criteria:

* Household member already participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2954 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-03-04 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of hospital admissions where the primary reason for admission is AECOPD | 12 months post randomisation
  A binary outcome assessing incidence of at least one AECOPD over 12 months after randomisation where patients needed hospitalisation (defined by hospital discharge letter/coding).

SECONDARY OUTCOMES:
Number of self-reported AECOPD every 3 months | 3, 6, 9 and 12 months post randomisation
  Self-reported AECOPD (including those for which admission is required) obtained by telephone calls
Number of Self-reported antibiotic and steroid prescriptions for AECOPD | 3, 6, 9 and 12 months post randomisation
  Self-reported number of hospitalisations due to AECOPD obtained by telephone calls
Number of all cause hospital admissions | 12 months post randomisation
  All cause hospital admission taken from Hospital Episode Statistics (HES) and/or participant self-report
Number of readmissions to hospital for AECOPD at 30 and 90 days | 12 months post randomisation
  Readmissions to hospital for AECOPD at 30 and 90 days taken from HES and/or participant self-report
Number of Bed days due to AECOPD | 12 months post randomisation
  Total in hospital bed days due to AECOPD taken from HES and/or participant self-report
Number of participant deaths from all causes | 12 months post randomisation
  All-cause mortality taken from HES and/or medical records
Number of unscheduled GP visits for AECOPD | 12 months post randomisation
  Self-reported unscheduled GP visits for AECOPD
Number of prescriptions for 2nd courses of antibiotics within 14 days of self-reported event (defined as treatment failure) | 12 months post randomisation
  Self-reported prescriptions for 2nd courses of antibiotics within 14 days of self-reported
Number of prescriptions for oral anti-fungals | 12 months post randomisation
  Self-reported prescriptions for oral anti-fungals (e.g. for oral thrush)
Quality of life by COPD assessment test | 3, 6, 9 and 12 months post randomisation
  Quality of life measured using the COPD assessment test (CAT) at 3 monthly intervals
Quality of life measured using the EuroQoL-5Dimension-5Level questionnaire | 3, 6, 9 and 12 months post randomisation
  Measured at 3 monthly intervals. The EQ-5D-5L generates a score from 5 to 25 (5 being 'no problem' on all of the 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression), the total score will be used for the economic evaluation only
Antibiotic resistance | at baseline, all AECOPD and 12 months post randomisation
  identification of antibiotic resistant pathogens within sputum culture
Healthcare resource utilisation | 3, 6 and 9 and 12 months post randomisation
  determined from participant self-report on bespoke questionnaire (in development)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Turner, Principal Investigator — The University of Birmingham and University Hospitals NHS Foundation Trust
Locations (1):
- West Midlands Clinical Research Network, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Datasets generated and analysed during the current study will be available upon request from Birmingham Clinical Trials Unit (BCTU: bctudatashare@contacts.bham.ac.uk). Data will typically be available within 6 months after the primary publication unless it is not possible to share the data. Only scientifically sound proposals from appropriately qualified Research Groups will be considered for data sharing. The request will be reviewed by the BCTU Data Sharing Committee in discussion with the CI and, where appropriate (or in absence of the CI) any of the following: the Trial Sponsor, the relevant Trial Management Group, and the independent Trial Steering Committee. A formal Data Sharing Agreement (DSA) may be required between respective organisations once the release of the data is approved and before data can be released. Data will be fully anonymised unless the DSA covers the transfer of patient identifiable information. Data transfer will use a secure and encrypted method.